CLINICAL TRIAL: NCT04003129
Title: Knowledge, Practice and Attitude of Paediatricians Regarding Early Childhood Caries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Ali Abd el-hafiez Hegazy, Principal Investigator, Cairo University
Other Study IDs: pediatricians and ECC
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Early Childhood Caries
Keywords: paediatrician; early childhood caries
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Data will be obtained through a written questionnaire for assessing knowledge, practice and attitude of paediatricians regarding early childhood caries.
  Data collected will be saved and tabulated on computer and finally statistically analysed.

SUMMARY:
To assess the knowledge, practice and attitude of paediatricians regarding early childhood caries and infant's oral health.

DETAILED DESCRIPTION:
According to The American Academy of Pediatric Dentistry, Early Childhood Caries ECC is defined as the presence of one or more decayed (noncavitated or cavitated lesions), missing (due to caries), or filled tooth surfaces in any primary tooth in a child under the age of six Early Childhood Caries is a serious oral health problem worldwide with a prevalence of 61.4% in preschool children in Egypt. Bottle-feeding during night-sleep, unhealthy diet with high sugar consumption, lack of parental awareness regarding their children oral health, low socioeconomic status and lack of access for dental care were all reported as risk factors for ECC .

ECC might lead to adverse effects on children's physical, psychological and social well-being, as the associated dental pain and tooth loss can negatively influence children's nutrition, phonetics, socializing and sleeping. Moreover, treating ECC represents a financial burden for both the family and health care organizations, as it usually necessitates the aid of general anaesthesia . Therefore, more attention and efforts should be made to obtain an early assessment of oral health status of infants and children and reach the high-risk groups of ECC within populations, in order to reduce the prevalence of ECC and consequently to improve the quality of life of these children .

Paediatricians are the first to contact the infants and their families and infants often have frequent and regular visits to them than to the dentists. Therefore the paediatricians have to recognize their role in the promotion of children's oral health by several means such as; assessing the child's risk of developing dental caries, providing basic screening services for early detection of dental problems, parental education, and referral of required conditions . This is in accordance to the American Academy of Paediatric Dentistry guidelines which recommends the utilization of different preventive strategies for the prevention and early detection of ECC and also emphasizes the importance of its initiation in the primary health care provider's. .

Gaining information about the knowledge, practice and attitude of paediatricians regarding early childhood caries and infant's oral health will help identifying the points of weakness and improving their knowledge which will facilitate the early assessment of the oral health status and delivery of preventive oral measures to the infants and children which in turn may reduce or even eliminate oral diseases.

ELIGIBILITY:
Inclusion Criteria:

* Paediatricians working in hospitals. Paediatricians treating infants and children less than 6 years.

Exclusion Criteria:

* Under graduate students and interns

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: paediatricians are doctors who treat childrens.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
knowledge, practice and attitude of paediatricians regarding early childhood caries | 1 year
  obtaining information about knowledge, practice and attitude of paediatricians regarding early childhood caries by questionnaire with a measuring unit binary and MCQ questions

REFERENCES:
- See also: Oral Health Status of Preschool Children in Egypt Hanaa — https://www.mendeley.com/catalogue/oral-health-status-preschool-children-egypt/
- See also: Policy on Early Childhood Caries (ECC): Classifications, Consequences, and Preventive Strategies — https://www.mendeley.com/catalogue/policy-early-childhood-caries-ecc-classifications-consequences-preventive-strategies-6/